CLINICAL TRIAL: NCT07110272
Title: The Impact of Pediatric Nurses' Hypothetical and Creative Reasoning Skills on the Provision of Quality Nursing Care: A Descriptive Study
Brief Title: How Pediatric Nurses' Reasoning Skills Affect Quality Nursing Care
Status: Not yet recruiting | Type: Observational
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, YAĞMUR ŞANCI, Asst. Prof. Dr., Fenerbahce University
Other Study IDs: 101.2024fbu
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Critical Thinking in Nursing; Pediatric Nursing Practice; Quality of Nursing Care; Clinical Reasoning
Keywords: Pediatric Nursing; Hypothetical Reasoning; Creative Reasoning; Nursing Care Quality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This descriptive study aims to examine the impact of pediatric nurses' hypothetical and creative reasoning skills on the quality of nursing care.

The research seeks to answer the following questions:

Do the sociodemographic characteristics of pediatric nurses influence the quality of nursing care they provide? Do pediatric nurses' hypothetical and creative reasoning skills affect the quality of the nursing care they deliver? Participants will be asked to select the response that best reflects their own perspective for each item. This process will take approximately 10 minutes.

DETAILED DESCRIPTION:
This study aims to investigate the relationship between pediatric nurses' hypothetical and creative reasoning skills and the quality of the nursing care they provide. The research is grounded in the premise that advanced cognitive reasoning capabilities are critical for delivering high-quality, patient-centered care in pediatric settings.

A descriptive, cross-sectional research design will be employed. The study population consists of pediatric nurses currently employed in various healthcare institutions across Turkey.

Data will be collected through a socio-demographic questionnaire, the Hypothetical and Creative Reasoning Scale for Nurses and the Quality of Nursing Care Scale. These tools will assess the nurses' cognitive reasoning skills and perceived nursing care quality.

Statistical analyses will be conducted to determine correlations between nurses' reasoning skills and the quality of care provided. This research will also explore whether socio-demographic characteristics (e.g., age, education level, years of experience) are associated with reasoning ability or care quality.

The findings are expected to contribute to the body of knowledge in nursing education and practice by emphasizing the importance of cognitive reasoning in nursing quality, particularly in pediatric settings.

ELIGIBILITY:
Inclusion Criteria:

* Currently working as a pediatric nurse during the time of the study

Exclusion Criteria:

* Not volunteering to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of the study will consist of pediatric nurses working in Türkiye, while the sample will include those who agree to participate in the research. The sampling method of the study has been determined as simple random sampling.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Do pediatric nurses' hypothetical and creative reasoning skills affect the quality of the nursing care they deliver? | August - September 2025
  It is hypothesized that higher scores in hypothetical and creative thinking skills among pediatric nurses will be associated with higher scores on the Quality of Nursing Care Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Fenerbahçe University, Ataşehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No